CLINICAL TRIAL: NCT06835491
Title: Prophylactic Anti-aRrhythmic Therapy With Amiodarone in Critically Ill Patients Admitted for an Out-of-hospital Cardiac Arrest With Initial Shockable Rhythm.
Acronym: PARACA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Hugo Bellut, Investigator coordonator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P23/08_PARACA
Record Dates: First submitted 2025-01-15; First posted 2025-02-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Ventricular Arrhythmias and Cardiac Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Amiodarone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amiodarone (Experimental): Initial loading dose of 300mg over 30 minutes in 250ml of glucose 5% solution. Continuous amiodarone infusion will be administered for 72 hours at a dose of 10 mg/kg without exceeding 900 mg/24h.
  Interventions: Drug: Amiodarone
- Control (No Intervention)

INTERVENTIONS:
Drug: Amiodarone — Initial loading dose of 300mg over 30 minutes in 250ml of glucose 5% solution. Continuous amiodarone infusion will be administered for 72 hours at a dose of 10 mg/kg without exceeding 900 mg/24h.
  Arms: Amiodarone

SUMMARY:
To determine if prophylactic administration of amiodarone for 72 hours in critically ill patients admitted after an OHCA with shockable rhythm, with a confirmed or a presumed cardiac cause, decreases the incidence of a composite endpoint of 30-day (starting from inclusion) all-cause mortality and/or severe in-hospital ventricular arrhythmia recurrence (ventricular fibrillation and/or ventricular tachycardia requiring intervention including re-arrest)

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥ 18 years
2. Admitted in intensive care unit
3. Out-of-hospital cardiac arrest with initial shockable rhythm
4. Presumed cardiac or unknown cause
5. Delay between ROSC and screening for randomisation < 6 hours
6. Informed consent from the patient or a surrogate or deferred consent
7. Affiliated to or benefiting from a social insurance

Exclusion Criteria:

1. Cardiac arrest secondary to an extra-cardiac cause (suspected or confirmed)
2. Indication for amiodarone decided by the physician at ICU admission
3. No central venous catheter available for continuous infusion of amidoarone
4. Thyroid disease under treatment
5. History of cardiac conduction disorders, not treated by permanent pacemaker
6. Any contra indication to amiodarone treatment
7. Refractory ventricular arrhythmia or electrical storm
8. Need for veno-arterial extracorporeal membrane oxygenation (VA-ECMO) at admission
9. Known limitations in therapy and Do Not Resuscitate-order
10. Moribund patient due to pre-arrest history (estimated life expectancy < 3 months)
11. Pregnant or breastfeeding women
12. Patient needing a nadolol treatment due to QT long syndrome or catecholaminergic polymorphic ventricular tachycardia
13. Patient with known pulmonary fibrosis
14. Patient with known interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 674 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Rate of Mortality and severe ventricular arrhythmia | 30 days
  The primary endpoint is a composite of 30-day (starting from inclusion) all-cause mortality and occurrence of severe in-hospital ventricular arrhythmia, defined by ventricular fibrillation and/or ventricular tachycardia requiring intervention occurring between inclusion and hospital discharge (or 30-day whichever the sooner).

SECONDARY OUTCOMES:
outcomes related with cardiac events | 90 days
  * Occurrence of ventricular fibrillation (VF)
  * Occurrence of ventricular tachycardia (VT) requiring or not intervention
  * Occurrence of atrial fibrillation (AF) and supraventricular tachycardia
  * Occurrence of cardiac re-arrest due to asystole
outcomes related with mortality | 90 days
  * ICU mortality
  * Hospital (and 30-day) mortality
  * Day 90 mortality
Duration of invasive mechanical ventilation | 90 days
Number of participants with outcomes related with amiodorane side effects | 5 days
  Number of the following side effects, patients could experimente (if applicable) during amiodarone infusion:
  * Conduction disorders
  * Hemodynamic consequences
  * Hepatic cytolysis
  * Anaphylaxis
Neurological outcome | 90 days
  M-Rankin scale (the lowest score is no handicap and the highest score is death) and Glasgow Outcome Score (the lowest score is the most severe coma)
Duration vasopressor infusion | 90 days
Length of ICU stay | 90 days
Length of stay in hospital | 90 days
Dose of the anti-arrhythmic drugs | 90 days
Number of days of anti-arrhythmic drugs | 90 days

CONTACTS AND LOCATIONS:
Locations (29):
- France (29):
  - Chu Amiens, Amiens
  - Chu Angers, Angers
  - CH annecy genevois, Annecy
  - Ch Argenteuil, Argenteuil
  - CH Mondor, Aurillac
  - CHU Brest, Brest
  - CH Brive, Brive-la-Gaillarde
  - Chu Caen, Caen
  - Chi Nord Ardennes, Charleville-Mézières
  - CHSF, Corbeil-Essonnes
  - CHD vendée, La Roche-sur-Yon
  - CH la rochelle, La Rochelle
  - Hcl, Lyon
  - Ap Hm, Marseille
  - Hopital Cartier, Massy
  - chi Gregoire, Montreuil
  - Hoptial Mulhouse, Mulhouse
  - CHU Nantes, Nantes
  - Clinique Ambroise Paré, Neuilly-sur-Seine
  - CHU Nice -MIR Archet, Nice
  - CHU Nice -MIR Pasteur, Nice
  - Chu Orléans, Orléans
  - CHU Cochin, Paris
  - Hopital saint joseph, Paris
  - CHU Poitiers, Poitiers
  - Chu Strasbourg, Strasbourg
  - CHI Toulon, Toulon
  - Chu Toulouse, Toulouse
  - CH Cotentin, Valognes

IPD SHARING:
Plan to Share IPD: No